CLINICAL TRIAL: NCT01014416
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Single Dose, Dose-escalation Study to Investigate the Safety, Tolerance, Pharmacokinetics and Pharmacodynamics of Tolvaptan in Healthy Korean Male Subjects Bipolar Disorder
Brief Title: Pharmacokinetics/Pharmacodynamics (PK/PD) Characteristics of Tolvaptan Tablet in Korean Healthy Male
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: SungWoo Hong, Korea Otsuka Pharmaceutical Co.,Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 156-KOA-0801
Record Dates: First submitted 2009-11-03; First posted 2009-11-17 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
Keywords: Healthy Korean male
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Single dose, Tolvaptan 15mg or Placebo/day
  Interventions: Drug: Tolvaptan 15mg or 30mg or 60mg or Placebo
- Arm 2 (Experimental): Single dose, Tolvaptan 30mg or Placebo/day
  Interventions: Drug: Tolvaptan 15mg or 30mg or 60mg or Placebo
- Arm 3 (Experimental): Single dose, Tolvaptan 60mg or Placebo/day
  Interventions: Drug: Tolvaptan 15mg or 30mg or 60mg or Placebo

INTERVENTIONS:
Drug: Tolvaptan 15mg or 30mg or 60mg or Placebo — Single dose of Tolvaptan 15mg or 30mg or 60mg or Placebo per day

SUMMARY:
To investigate the safety, tolerance, pharmacokinetics and pharmacodynamics of tolvaptan 15, 30 and 60 mg after single oral administration in healthy Korean male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Korean male subjects between 20 and 45 years of age, inclusive.
2. Body Mass Index (BMI) of 20 to 26 kg/m2, body,weight ≥ 50kg BMI = weight (kg)/height2(m)
3. Informed consent from the subjects

Exclusion Criteria:

1. Clinically significant abnormality of respiratory, cardiovascular, hepatic, neurologic, endocrine, hematologic, urinary, psychiatric.
2. History of gastrointestinal disease or surgery which can affect intestinal absorption of the study drug.
3. History of any significant drug allergy or hypersensitivity.
4. AST or ALT > 1.25 times upper normal limit at screening clinical laboratory test
5. Supine blood pressure after resting for ≥ 3 minutes, higher than 140/90 mmHg or lower than 100/50 mmHg, Supine pulse, after resting for ≥ 3 minutes, outside the range of 40 to 90 beats/minute.
6. Subjects who had history of drug abuse or alcohol addiction
7. Subjects who used of any prescription drug or herbal medication within 2 weeks prior to the first dosing of the study drug, or any over-the-counter or vitamin supplements within 1 week prior to the first dosing (However, investigators can judge the subject, who has taken the medications during those periods above, eligible for the trial if all other conditions are satisfied)
8. The investigator judges the subject not eligible for the study after reviewing clinical laboratory results or other reasons.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
PK parameters: AUC, Cmax, Tmax | 1 day
PD parameters: 24 hour fluid balance | 1 day
Safety: adverse event, body weight, physical examination, vital sign, ECG, clinical laboratory test | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea